CLINICAL TRIAL: NCT02133794
Title: Tomosynthesis Use in Detecting Subtle Occult Hip Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical Imaging Informatics Research Centre at McMaster (Other)
Responsible Party: Principal Investigator, Naveen Parasu, Dr. Naveen Parasu, Medical Imaging Informatics Research Centre at McMaster
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Parasu-001
Record Dates: First submitted 2014-04-23; First posted 2014-05-08 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-04

CONDITIONS: Hip Fracture
Keywords: Hip fracture; Tomosynthesis; X-ray; Emergency room
MeSH Terms: conditions — Hip Fractures; Emergencies | interventions — Mammography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tomosynthesis (Experimental)
  Interventions: Device: Tomosynthesis

INTERVENTIONS:
Device: Tomosynthesis
  Other Names: GE Discovery 650

SUMMARY:
The purpose of this project is to determine if using tomosynthesis, in conjunction with x-ray, is better at detecting hip fractures than using x-ray alone. The goal of this study will be to include the use of tomosynthesis with x-ray as usual practice when a patient comes to the emergency room with symptoms of a hip fracture.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged > 18 years who/se:
* Present at the ER with a possible hip fracture and
* Have a negative x-ray for a hip fracture
* Physician has a high clinical suspicion of a hip fracture
* Provide provision of informed consent

Exclusion Criteria:

* Hip prosthesis on the same side of the suspected hip fracture
* Other serious medical illness that is likely to interfere with study participation
* Significant psychiatric illness, senility, dementia, alcohol or substance abuse, which could impair the ability to provide informed consent and to adhere to the trial procedures
* Pregnant or suspected pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with hip fracture detected with tomosynthesis versus x-ray alone. | Participants will be followed up to 3 months post tomosynthesis exam.

SECONDARY OUTCOMES:
ER wait time | End of study

CONTACTS AND LOCATIONS:
Locations (1):
- Juravinski Hospital, Hamilton, Ontario, Canada